CLINICAL TRIAL: NCT02480166
Title: Comparative Efficacy of Fixed-dose Combination of Sofosbuvir and Ledipasvir for 8 or 12 Weeks for Chronic Hepatitis C Genotype 6
Brief Title: Comparative Efficacy of Fixed-dose Combination Sofosbuvir + Ledipasvir, 8 vs. 12 Weeks in Chronic Hepatitis C Genotype 6
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Mindie H. Nguyen, Associate Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33196
Record Dates: First submitted 2015-06-17; First posted 2015-06-24 (Estimated); Results first posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-08

CONDITIONS: PT-NANBH
Keywords: hepatitis C, genotype 6
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 8 weeks SOF/LED (Experimental): Patients that are treatment naïve and without cirrhosis will be assigned to 8 weeks of treatment with fixed-dose combination sofosbuvir (400 mg) and ledipasvir (90 mg) daily.
  Interventions: Drug: 8 weeks SOF/LED
- 12 weeks SOF/LED (Experimental): Patients that are either treatment experienced or are cirrhotic will be assigned to 12 weeks of treatment with fixed-dose combination sofosbuvir (400 mg) and ledipasvir (90 mg) daily.
  Interventions: Drug: 12 weeks SOF/LED

INTERVENTIONS:
Drug: 8 weeks SOF/LED — Eligible and consenting patients will be treated with sofosbuvir 400 mg daily and ledipasvir 90 mg daily for 8 weeks. Patients that are treatment naïve and without cirrhosis will be assigned to 8 weeks of treatment. The drug will be administered orally, per manufacturers' instructions, and can be taken with or without food.
  Other Names: Harvoni; Solvaldi
  Arms: 8 weeks SOF/LED
Drug: 12 weeks SOF/LED — Eligible and consenting patients will be treated with sofosbuvir 400 mg daily and ledipasvir 90 mg daily for 8 weeks. Patients that are not treatment naïve or have cirrhosis will be assigned to 12 weeks of treatment. The drug will be administered orally, per manufacturers' instructions, and can be taken with or without food.
  Other Names: Harvoni; Solvaldi
  Arms: 12 weeks SOF/LED

SUMMARY:
The primary objectives of this study are to describe the efficacy of:

1. 8-week treatment of SOF/LED for treatment-naïve, non-cirrhotic, HCV genotype 6
2. 12-week treatment of SOF/LED for all other HCV-6 populations

DETAILED DESCRIPTION:
The secondary objective of this study is to describe safety, persistency, and tolerability of SOF/LED in patients with HCV-6.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18 years
2. HCV genotype 6 or indeterminate and later assessed at Screening and confirmed as genotype 6
3. Selected to start on treatment by their treating providers
4. Willing and able to provide informed consent
5. Able to comply with dosing instructions for study drug administration and able to complete the study schedule of assessments
6. Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative pregnancy test on Baseline
7. Male subjects and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception
8. Lactating females must agree to discontinue nursing before the study drug is administered

Exclusion Criteria:

1. Previous recipient of a liver transplant
2. Co-infection with human immunodeficiency virus (HIV) or hepatitis B (HBV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mindie H Nguyen, MD, MAS, Principal Investigator — Stanford University
Locations (4):
- United States (4):
  - Stanford University Medical Center, Palo Alto, California
  - San Jose Gastroenterology, San Jose, California
  - Liver and Digestive Consultants, Houston, Texas
  - Digestive Health Associates, Plano, Texas

REFERENCES:
- [Background] Lawitz E, Gane EJ. Sofosbuvir for previously untreated chronic hepatitis C infection. N Engl J Med. 2013 Aug 15;369(7):678-9. doi: 10.1056/NEJMc1307641. No abstract available. PMID 23944316
- [Background] Lam KD, Trinh HN, Do ST, Nguyen TT, Garcia RT, Nguyen T, Phan QQ, Nguyen HA, Nguyen KK, Nguyen LH, Nguyen MH. Randomized controlled trial of pegylated interferon-alfa 2a and ribavirin in treatment-naive chronic hepatitis C genotype 6. Hepatology. 2010 Nov;52(5):1573-80. doi: 10.1002/hep.23889. PMID 21038410
- [Background] Afdhal N, Reddy KR, Nelson DR, Lawitz E, Gordon SC, Schiff E, Nahass R, Ghalib R, Gitlin N, Herring R, Lalezari J, Younes ZH, Pockros PJ, Di Bisceglie AM, Arora S, Subramanian GM, Zhu Y, Dvory-Sobol H, Yang JC, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Sulkowski M, Kwo P; ION-2 Investigators. Ledipasvir and sofosbuvir for previously treated HCV genotype 1 infection. N Engl J Med. 2014 Apr 17;370(16):1483-93. doi: 10.1056/NEJMoa1316366. Epub 2014 Apr 11. PMID 24725238
- [Background] Afdhal N, Zeuzem S, Kwo P, Chojkier M, Gitlin N, Puoti M, Romero-Gomez M, Zarski JP, Agarwal K, Buggisch P, Foster GR, Brau N, Buti M, Jacobson IM, Subramanian GM, Ding X, Mo H, Yang JC, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Mangia A, Marcellin P; ION-1 Investigators. Ledipasvir and sofosbuvir for untreated HCV genotype 1 infection. N Engl J Med. 2014 May 15;370(20):1889-98. doi: 10.1056/NEJMoa1402454. Epub 2014 Apr 11. PMID 24725239
- [Background] Chao DT, Abe K, Nguyen MH. Systematic review: epidemiology of hepatitis C genotype 6 and its management. Aliment Pharmacol Ther. 2011 Aug;34(3):286-96. doi: 10.1111/j.1365-2036.2011.04714.x. Epub 2011 May 29. PMID 21623850

RESULTS

PARTICIPANT FLOW:
Groups:
- Extended Treatment to 12 Weeks SOF/LED: Subjects without cirrhosis or prior treatment history received extended treatment to 12 weeks by investigator's preference
Period: Overall Study
Arm/Group | 8 Weeks SOF/LED | 12 Weeks SOF/LED | Extended Treatment to 12 Weeks SOF/LED
Started | 20 | 36 | 4
Completed | 20 | 36 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 8 Weeks SOF/LED | 12 Weeks SOF/LED | Extended Treatment to 12 Weeks SOF/LED | Total
Number analyzed (Participants) | 20 | 36 | 4 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (8) | 60 (12) | 54 (10) | 59 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 1 | 25
  Male | 11 | 21 | 3 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Vietnamese | 16 | 30 | 4 | 50
  Cambodian | 1 | 3 | 0 | 4
  Other Asian | 3 | 3 | 0 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 36 | 4 | 60
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.4 (4.2) | 24.2 (2.7) | 24.1 (3.6) | 23.6 (3.3)
Comorbidities [Count of Participants; unit: Participants]
  Diabetes | 1 | 6 | 0 | 7
  Hypertension | 5 | 10 | 0 | 15
  Hyperlipidemia | 3 | 6 | 0 | 9
  Coronary Artery Disease (CAD) | 0 | 1 | 0 | 1
  Chronic Obstructive Pulmonary Disease (COPD) | 0 | 1 | 0 | 1
HCV Genotype SubType [Count of Participants; unit: Participants]
  a/b | 2 | 9 | 2 | 13
  c-l | 8 | 15 | 2 | 25
  c | 1 | 0 | 0 | 1
  m | 0 | 2 | 0 | 2
Baseline Cirrhosis [Count of Participants; unit: Participants] | 0 | 27 | 0 | 27
Decompensated Cirrhosis [Count of Participants; unit: Participants] — Decompensated cirrhosis is defined as presence/history of variceal bleeding, hepatic encephalopathy, or ascites at baseline.
  Participants | 0 | 2 | 0 | 2
Hepatocellular Carcinoma [Count of Participants; unit: Participants] | 0 | 3 | 0 | 3
Prior Treatment [Count of Participants; unit: Participants] | 0 | 15 | 0 | 15
Proton Pump Inhibitor (PPI) usage [Count of Participants; unit: Participants] | 3 | 9 | 0 | 12
MELD, cirrhotics only [Mean (Standard Deviation); unit: units on a scale] — The Model for End-Stage Liver Disease (MELD) Score uses the patient's values for serum bilirubin, serum creatinine, and the international normalized ratio for prothrombin time (INR) to predict survival. It is calculated according to the following formula: MELD = 3.78×ln[serum bilirubin (mg/dL)] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43. The total possible range for MELD scores is 6 (less ill) to 40 (gravely ill).
  units on a scale | 0 (0) | 6.9 (1.6) | 0 (0) | 6.9 (1.6)
log10 HCV RNA [Mean (Standard Deviation); unit: log10 (IU/ml)] | 6.2 (0.8) | 6.5 (0.6) | 7.2 (0.3) | 6.5 (0.7)
White Blood Cell Count (WBC) [Mean (Standard Deviation); unit: K/uL] | 5.5 (1.4) | 6.0 (2.1) | 5.3 (0.5) | 5.8 (1.8)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 14.3 (1.3) | 14.2 (1.6) | 14.8 (1.1) | 14.2 (1.5)
Platelets [Median (Inter-Quartile Range); unit: K/uL] | 213 [186 to 240] | 181 [133 to 223] | 201 [189 to 225] | 201 [151 to 223]
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.8 (0.1) | 0.9 (0.2) | 0.9 (0.1) | 0.8 (0.2)
International Normalized Ratio (INR) [Mean (Standard Deviation); unit: ratio] — The INR is based on the ratio of the patient's prothrombin time and the normal mean prothrombin time. The normal range for a healthy person who is not on anticoagulant therapy is 0.8-1.2, while higher values are targeted for people on anticoagulant therapy.
  ratio | 1.0 (0.2) | 1.0 (0.1) | 1.0 (0.0) | 1.0 (0.1)
Total bilirubin [Mean (Standard Deviation); unit: mg/dL] | 0.7 (0.1) | 0.8 (0.4) | 0.9 (0.1) | 0.7 (0.3)
Aspartate Aminotransferase (AST) [Median (Inter-Quartile Range); unit: U/L] — AST is an enzyme that is secreted from the liver and can be found in liver, heart, muscle tissue, pancreas and kidneys. Elevated levels of AST may indicate inflammation or liver damage. Normal range for AST is typically 10-40 U/L.
  U/L | 36 [27 to 44] | 48 [33 to 95] | 28 [21 to 34] | 39 [29 to 69]
Alanine Aminotransferase (ALT) [Median (Inter-Quartile Range); unit: U/L] — ALT is an enzyme that is secreted by the liver into the blood. Main storage of this enzyme is in the liver and elevated levels of ALT in the blood may indicate liver inflammation or damage. Normal range for ALT is typically between 7-56 U/L.
  U/L | 44 [31 to 59] | 68 [46 to 105] | 33 [21 to 41] | 59 [36 to 76]
Albumin [Mean (Standard Deviation); unit: g/dL] | 4.3 (0.4) | 4.0 (0.7) | 3.5 (1.5) | 4.0 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Sustained Virologic Response (SVR) log10 HCV RNA PCR <25 IU/mL 12 Weeks Post-treatment
Time Frame: 12 weeks after end of therapy
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Extension to 12 Weeks SOF/LED: Subjects without cirrhosis or prior treatment history received extended treatment to 12 weeks by investigator's preference
Arm/Group | 8 Weeks SOF/LED | 12 Weeks SOF/LED | Treatment Extension to 12 Weeks SOF/LED
Number analyzed (Participants) | 20 | 36 | 4
Participants | 19 | 34 | 4

2. Secondary Outcome: Number of Participants Who Experienced Serious Adverse Events (SAEs) and/or Adverse Events (AEs) From Informed Consent to 12 Weeks Post-treatment.
Description: Adverse events were defined using Common Terminology Criteria for Adverse Events v3.0 (CTCAE)
Time Frame: Day 1 of treatment to 12 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 8 Weeks SOF/LED | 12 Weeks SOF/LED | Extended Treatment to 12 Weeks SOF/LED
Number analyzed (Participants) | 20 | 36 | 4
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For each subject, AEs and SAEs are recorded after informed consent is obtained until 12 weeks post treatment.
Description: A Serious Adverse event must be reported if it occurs during a subject's participation in the Study (whether receiving Study Product or not) and within 30 days of receiving the last dose of Study Product.
  Any serious adverse event that is ongoing when a subject completes his/her participation in the Study must be followed until the event resolves or stabilizes, returns baseline condition, or can be attributed to agents(s) other than the Study Product, or unrelated to Study conduct.
Arm/Group | 8 Weeks SOF/LED | 12 Weeks SOF/LED | Extended Treatment to 12 Weeks SOF/LED
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/36 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/20 | 2/36 | 0/4
Other Adverse Events (participants affected / at risk) | 2/20 | 5/36 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 Weeks SOF/LED (N=20) | 12 Weeks SOF/LED (N=36) | Extended Treatment to 12 Weeks SOF/LED (N=4)
Upper GI Bleed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — H.pylori-related bleeding gastric ulcer unrelated to study treatment. Subject achieved SVR 12.
Surgical correction of left wrist fracture (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — Surgical correction for wrist fracture due to a mechanical fall unrelated to study treatment. Subject achieved SVR 12.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 Weeks SOF/LED (N=20) | 12 Weeks SOF/LED (N=36) | Extended Treatment to 12 Weeks SOF/LED (N=4)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0) — Fatigue
Insomnia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (General disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Our population was small and our study was not powered to be able to determine significant differences between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No